CLINICAL TRIAL: NCT03021421
Title: The Effect of Unilateral Spinal Anaesthesia and Psoas Compartment With Sciatic Block on the Postoperative Pain Management in Total Knee Artroplastic Surgery
Brief Title: Comparison of Two Regional Technics In Knee Artroplasty
Acronym: CTRTIKA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Ebru Canakci, M.D, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OrduU
Record Dates: First submitted 2016-02-19; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Analgesia; Anesthesia; Functional
Keywords: Total knee arthroplasty; unilateral spinal anaesthesia; psoas compartment block; sciatic nerve block; haemodynamic effects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group USA (Sham Comparator): (Marcain Heavy 0.5%; AstraZeneca®, London, UK) using a 25-G Quincke spinal injector (B. Braun®, Melsungen, Germany).
  Interventions: Procedure: intratechal (subarachnoidal )injection
- Group PCS (Active Comparator): (Stimupleks A; B. Braun®, Melsungen AG, Germany) to lumbar plexus in psoas muscle compartment (injected material 20 ml local anaesthetic mixture5 ml of 2% lidocaine + 15 ml of 0.5% bupivacaine)
  %2 Aritmal ampul (Osel İlaç,Turkey) and Marcaine %0.5 flacon (AstraZeneca®, London, UK)
  Interventions: Procedure: lombar plexus and sciatic nerve injection

INTERVENTIONS:
Procedure: intratechal (subarachnoidal )injection — 10 mg (2 cc) intrathecal single shot injection
  Other Names: Marcaine Spinal 0,5 % Heavy ampule
  Arms: Group USA
Procedure: lombar plexus and sciatic nerve injection — USG -guided lumbar plexus visualised and 20 ml local anaesthetic mixture (15 cc %0,5 Bupivacaine Hydrochloride 5 cc and %2 Lidocaine 5 cc ) for lombar plexus single shot injection
  Other Names: Marcaine %0,5 20 cc flacon and Aritmal %2 ampule
  Arms: Group PCS

SUMMARY:
Purpose: This prospective, randomised, controlled, single-blind, multicentre study was designed to investigate the effects of peripheral nerve block methods (applied using unilateral spinal anaesthesia [USA] on elderly patients scheduled to undergo total knee arthroplasty) on perioperative haemodynamic parameters and the postoperative analgesia period.

Materials and Methods: Sixty patients in the American Society of Anesthesiologists (ASA) Physical Status II-III group were randomly divided into two groups. Spinal anaesthesia was performed in the USA group, in the lateral position through the intervertebral space, with 2 ml of hyperbaric bupivacaine (L4-L5 or L3-L4); 0.5% bupivacaine hydrochloride and 2% lidocaine were combined for the psoas compartment-sciatic (PCS) group, and the mixture was used for psoas compartment block (PCB) and sciatic nerve block. The haemodynamic parameters were recorded every 5 minutes until the end of the preoperative and perioperative operation periods and postoperative first analgesic application time.

DETAILED DESCRIPTION:
In this prospective, randomised, multicentric and single-blind study, 60 patients who were diagnosed with gonarthrosis in the outpatient clinic of Ordu University Training Hospital and Ordu State Hospital between January 1, 2015 and June 30, 2015, and planned for total knee arthroplasty, were included. Patients who were allergic to local anaesthetics, had neurological disease, had infections in the intervention area, did not cooperate, or did not agree to the intervention were excluded from the study. After receiving informed consent from the patients, they were divided into two groups using the closed envelope method: the USA Group was the spinal anaesthesia (SA) group (n = 30), and the PCS group was the PCB and sciatic nerve block group (n = 30). All of the patients planned for surgery were monitored in terms of non-invasive arterial blood pressure, heart rate (HR) and peripheral haemoglobin oxygen saturation (SpO2). Peripheral vascular access was established using an 18-G cannula before the block operation, and 500 ml of 0.9% NaCl solution was infused for 20 minutes followed by the intravenous administration of 0.07 mg/kg midazolam (Dormicum®; Roche, Basel, Switzerland). The haemodynamic parameters were recorded every 5 minutes until the end of the preoperative and perioperative operation period. Next, 2 ml of hyperbaric bupivacaine hydrochloride (Marcain Heavy 0.5%; AstraZeneca®, London, UK) was administered to patients in the USA group in the lateral decubitus position, after regional sterilisation, through the selected intervertebral space (L4-L5 or L3-L4) using a 25-G Quincke spinal injector (B. Braun®, Melsungen, Germany). After remaining in this position for 15 minutes after the procedure, the patients were changed to the supine position. Patients in the PCS group were changed to the lateral decubitus (Simms) position. Following the sterilisation and covering procedures required for blockade of the lumbar plexus somatic nerves, the abdominal settings were selected on the ultrasound device (Mindray DC-T6 VET®, Shenzhen, China). The depth was set at 11-12 cm, and the frequency was set at 4-8 MHz. A convex ultrasonography (USG) probe was placed 4 cm laterally on the middle line at the L3-L5 level. The transverse process was longitudinally identified using an USG probe. The 'trident sign' (three-pronged spear appearance) acoustic shadow of the transverse process is characteristic. After viewing the psoas muscle at the depth of the transverse process, the needle was inserted using an out-plane approach. While using a nerve stimulator simultaneously (Stimupleks A; B. Braun®, Melsungen AG, Germany), the stimulation current was reduced to the 0.5-1.0 mA level when contraction of the quadriceps muscle was observed, and 20 ml of local anaesthetic (5 ml of 2% lidocaine + 15 ml of 0.5% bupivacaine) was injected. The local anaesthetic was observed to disperse around the lumbar plexus with USG. Sciatic nerve block was applied as follows: the patients' positions were not changed, and the skin was disinfected in the same position (lateral decubitus position). Following the required covering process, the USG settings were applied for optimum visualisation. The depth was set as 3-6 cm, and frequency as 2-8 MHz. The convex USG probe was placed in the subgluteal area in the transverse position. After determining the sciatic nerve, the injector was inserted into the lateral edge of the probe as in-plane and proceeded towards the nerve. When using the nerve stimulator simultaneously (Stimupleks A; B. Braun®), the stimulation current was reduced to 0.2-0.5 mA until contractions became visible. The local anaesthetic was observed to disperse around the sciatic nerve with USG by administering 20 ml of local anaesthetic (5 ml of 2% lidocaine + 15 ml of 0.5% bupivacaine) following negative aspiration with the injector. The patients were changed to the supine position. Surgery was allowed when effective sensory block reached with at least a T10 dermatome.

After the procedure, the patients were changed to the supine position. The application times of both techniques were recorded as the technique application times. While the analgesia level was evaluated using the pinprick test, the degree of motor block was assessed using the modified Bromage scale (0: no block, 1: hip flexion is blocked when the knee is extended, 2: knee flexion is blocked, 3: full motor block). Additionally, the sensory and motor blocks were evaluated at 5-minute intervals using the measurements of the haemodynamic parameters after the administration of medications. No case was excluded from the study because of block failure; thus, the data of all the cases in both groups were analysed.

Surgical intervention was initiated after the development of a full motor block. The time from the beginning of surgical incision until the completion of the procedure was recorded as the operation period. A decrease in the mean basal arterial pressure of 25% or more was considered as hypotension; in this case, ephedrine was administered as 5 mg intravenously (i.v.), and 5 ml/kg additional crystalloid fluid was given. Heart rates less than 50 beats/minute were considered as bradycardia, and atropine was administered as 0.5 mg i.v. All of the patients were administered 3 l/minute O2 through the mask and 5 ml/kg/hour maintenance crystalloid i.v. fluid during the surgery. The motor block return time and first analgesic requirement time were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Between 50-80 age patients who have gonarthrosis

Exclusion Criteria:

* under 50 year
* above 80 years
* and who have local anaesthetic allergy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Postoperative VAS values | postoperative first 24 hour
  Visual Analog Scale (mm)

SECONDARY OUTCOMES:
Perioperative Heart Rate | perioperative 150 minute
  Beat to beat variability
Perioperative Mean Arterial Pressure | perioperative 150 minute
  mmHg

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Canakci E, Unal D, Guzel Y. The Effect of Unilateral Spinal Anaesthesia and Psoas Compartment with Sciatic Block on the Postoperative Pain Management in Total Knee Artroplastic Surgery. Pain Res Manag. 2017;2017:4127424. doi: 10.1155/2017/4127424. Epub 2017 Jan 31. PMID 28255259